CLINICAL TRIAL: NCT03085004
Title: CHARM II: Chemotherapy for Ablation and Resolution of Mucinous Pancreatic Cysts: a Prospective, Randomized, Double-blind, Multi-center Clinical Trial
Brief Title: CHARM II: Chemotherapy for Ablation and Resolution of Mucinous Pancreatic Cysts
Acronym: CHARM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matthew T. Moyer, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5206; 1R01CA222648 (NIH)
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cyst; EUS-FNA
Keywords: Pancreatic cyst; EUS-FNA; Chemotherapy; Endoscopic ultrasound-guided fine needle infusion; paclitaxel; gemcitabine; cyst ablation
MeSH Terms: conditions — Pancreatic Cyst | interventions — Ethanol; Saline Solution; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Cyst will be lavaged for 3 to 5 minutes with >/=99% ethanol. Following lavage with >/=99% ethanol, the cyst will be infused with an admixture of (3mg/ml paclitaxel + 19mg/ml gemcitabine).
  Interventions: Drug: Ethanol; Drug: Paclitaxel + Gemcitabine admixture
- Study group (Experimental): Cyst will be lavaged for 3 to 5 minutes with normal saline. Following lavage with normal saline, the cyst will be infused with an admixture of (3mg/ml paclitaxel + 19mg/ml gemcitabine).
  Interventions: Drug: Normal saline; Drug: Paclitaxel + Gemcitabine admixture

INTERVENTIONS:
Drug: Ethanol — The cyst will be lavaged for 3 to 5 minutes using >/=99% ethanol as the lavage agent prior to infusing the cyst with the paclitaxel + gemcitabine admixture.
  Arms: Control Group
Drug: Normal saline — The cyst will be lavaged for 3 to 5 minutes using normal saline as the lavage agent prior to infusing the cyst with the paclitaxel + gemcitabine admixture.
  Arms: Study group
Drug: Paclitaxel + Gemcitabine admixture — Following lavage, cysts will be infused with an admixture of 3mg/ml paclitaxel and 19mg/ml gemcitabine.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of chemotherapeutic pancreatic cyst ablation using ethanol lavage followed by the infusion of a dual-agent chemotherapeutic cocktail (paclitaxel + gemcitabine) compared with alcohol-free saline lavage followed by infusion of the same dual-agent chemotherapeutic cocktail (paclitaxel + gemcitabine) for the ablation of pancreatic cystic neoplasms using endoscopic ultrasound guided fine needle infusion (EUS-FNI) for agent delivery.

DETAILED DESCRIPTION:
Pancreatic cystic lesions are increasingly encountered and typically discovered incidentally on cross-sectional imaging, occurring in approximately 2% of all American adults with a 37% prevalence in individuals over 80. Most of these cysts are mucinous (neoplastic) in origin and represent precursor lesions for pancreatic adenocarcinoma.

Discovering a pancreatic cyst typically presents a treatment dilemma, with options including either indefinite radiographic surveillance with MR (magnetic resonance) or CT imaging or surgical resection, both of which have significant limitations. Surveillance carries significant economic and possible psychological burdens while waiting for signs of malignancy to develop, as well as radiation exposure with computed tomography. On the other hand, surgical resection possesses a significant risk of serious adverse events (20%-40%) and mortality (1-2%). This clinical dilemma delineates the pressing need to develop effective, but more minimally invasive approaches for the elimination of these premalignant pancreatic cysts, and among these, endoscopic ultrasound guided fine needle infusion (EUS-FNI) has emerged as an innovative and promising approach. Between November 2011 and December 30, 2015, investigators from interventional endoscopy, surgical oncology, hematology oncology, and pathology of the Penn State Hershey Medical Center conducted the CHARM I clinical trial. This was a prospective, randomized, double-blind, single-center study with an N of 46 patients required for 80% power to prove non-inferiority. Final results from CHARM I were as follows: Patients treated included 23 females and 16 males with the majority of lesions located in the body and head of the pancreas. Both the alcohol and alcohol-free groups recorded a 47% rate of complete ablation at 6 months, which increased to 64% for both groups at the 1 year follow-up. One subject experienced a complication in the alcohol arm (6%), and no subjects experienced complications in the alcohol-free arm.

The overall objectives of CHARM II are to verify the significant findings of CHARM I in a multi-center clinical trial as requested by national investigators in this field. We expect that administering a specifically designed chemotherapeutic cocktail without prior ethanol lavage will result in an equivalent rate of cyst resolution with fewer complications when compared with lavage using alcohol. The results of this study will provide important information about the most efficient and safest method for treating premalignant pancreatic cysts, an important step for treating these lesions with a minimally invasive technique and preventing their progression to pancreatic cancer. Standard alternative treatment options for this patient group (if not taking part in this study) would be ongoing periodic radiographic surveillance with MR or CT imaging waiting for signs of malignancy to develop or to consider surgical resection (an option with significant rates of morbidity and mortality).

This is an investigator-initiated, prospective, randomized, double-blinded, multi-center study evaluating ethanol lavage and chemotherapy for the ablation of mucinous and indeterminate type pancreatic cysts with malignant potential. Participants will be screened for the study according to inclusion and exclusion criteria. After confirming their eligibility, patients will be randomized to one of the following EUS-FNI treatment arms in a 1:1 ratio:

Control arm: After removal of cyst fluid, cysts will be lavaged for 3 to 5 minutes with >/=99% ethanol and then infused with an admixture of 3 mg/ml paclitaxel and 19 mg/ml gemcitabine.

Experimental arm: After removal of cyst fluid, cysts will be lavaged for 3 to 5 minutes with normal saline and then infused with an admixture of 3 mg/ml paclitaxel and 19 mg/ml gemcitabine.

Patients will be contacted by the study team via phone call at both 72 hours and 30 days after their EUS procedure to assess any adverse events that may have occurred. Within 2-3 weeks of the having the EUS procedure, patients will receive the cyst fluid pathology results. At 3 months after the initial procedure, patients will undergo a follow-up EUS examination in the same manner as the initial EUS exam. During this exam, a complete pancreaticobiliary evaluation will be conducted, and the diameter of the previously treated cyst will be measured in the x and y dimensions to assess the 3 month response. Any cyst still >15mm and amenable to repeat ablation will undergo a second EUS-guided chemoablation treatment using the same lavage that the patient was randomized to initially. At both 12 months and 24 months after the initial procedure, the patient will be seen in the GI clinic and undergo either an MRI-MRCP (magnetic resonance cholangiopancreatography) or enhanced CT scan for a full pancreaticobiliary evaluation to assess the end-point treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects over the age of 18.
* Patients with a previously-detected pancreatic cyst(s) 2-5 cm in diameter which is consistent with a mucinous type cyst as per ASGE guidelines, including indeterminate type cysts.
* Able to give written informed consent.
* Capable of safely undergoing endoscopy with deep sedation or general anesthesia.

Exclusion Criteria:

* Lesions which are consistent with a benign cyst by clinical, cytological, chemical, and radiographic evaluation as per ASGE guidelines (i.e., consistent with a pseudocyst or serous cystadenoma).
* Known or suspected pancreatic cancer or pathologic lymphadenopathy.
* Cysts with the following high-risk features: main pancreatic duct dilation of > 5mm, epithelial type mural nodules (> 2mm)33, pathologically thick wall/septation (> 2mm), cytology showing high grade dysplasia or "suspicious for malignancy", signs of common bile duct or pancreatic duct obstruction, solid mass component within or associated with the cyst (> 2mm), pancreatic duct stricture associated with tail atrophy, or previous fine needle aspiration failure due to excessive cyst fluid viscosity. (Of note, the following higher-risk features ARE eligible: recent growth in size, atypical cells on cytology, and symptoms referable to the pancreas.)
* Septated cysts with > 4 compartments.
* Confirmed acute pancreatitis within the last 6 months.
* Baseline lab values (must be within 6 months of consent date) in the following ranges: white blood cells > 14 or < 2 K/uL, hematocrit <30%, platelets <30 K/uL, non-pharmacologic INR >1.7, CA19-9 >2x ULN, lipase >2x ULN, creatinine >3.0 mg/dl (unless stable on renal replacement therapy), ALT >500 U/L, total bilirubin >2.5 mg/dl.
* Any pre-existing or discovered medical condition that would, at the discretion of the investigator, interfere with the completion of and/or participation in the existing protocol. This includes severe pre-existing medical conditions which would preclude a reasonable 5 year life expectancy (and thus neutralize the patient's benefit from ablating a premalignant type pancreatic cyst).
* Pregnancy, breastfeeding, or incarcerated individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving complete cyst resolution at 12 months | 12 months post initial treatment
  This is defined as Complete response greater than or equal to 95% reduction in cyst volume and measured by "r" as cyst volume 4/3×π×r3 at 12 months post initial treatment
Percentage of subjects achieving complete cyst resolution at 24 months of long term follow up | 24 months post initial treatment
  This is defined as Complete response greater than or equal to 95% reduction in cyst volume and measured by "r" as cyst volume 4/3×π×r3 at 24 months post initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Moyer, MD, MS, Principal Investigator — Penn State Health Milton S Hershey Medical Center
Locations (2):
- United States (2):
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No